CLINICAL TRIAL: NCT03571399
Title: Mortality and Morbidity in a Large Cohort of Asplenic Patients: a Nationwide Survey From the Italian Network on Asplenia
Brief Title: A Nationwide Italian Survey on Asplenia
Status: Completed | Type: Observational
Sponsor: Società Italiana Talassemie ed Emoglobinopatie (Other)
Collaborators: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Sponsor
Other Study IDs: Asplenia
Record Dates: First submitted 2018-06-07; First posted 2018-06-27 (Actual); Last update posted 2018-06-28 (Actual); Status verified 2018-05

CONDITIONS: Splenectomy; Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Spleen is involved in several functions, such as the production of protective antibodies, the removal of unwanted particulate matter from the blood (eg bacteria) and also the storing of blood cells, especially white cells and platelets. Asplenia is a status due to spleen absence or dysfunction, which results from several rare diseases. Congenital Asplenia is a condition with absent or dysfunctional spleen, associated with other congenital abnormalities; functional asplenia is a status with present but dysfunctional spleen, related to many rare diseases, such as sickle cell disease, thalassemia, essential thrombocythaemia, lymphoproliferative diseases and splenectomy is the surgical removal of the spleen in order to treat a huge number of rare hematological and oncological diseases. So, asplenia is the final result of a numerous variety of rare disorders, and it leads to a high risk of infections and thrombotic events with significant mortality and morbidity. Antibiotic prophylaxis and specific vaccinations are recommended in this high risk population but adherence was shown to be very poor. A national register was demonstrated to improve population outcomes and reduce health care costs and facilitate research and public health purposes in this target population. In Europe very little experience exists in comprehensive national program for management of asplenia, and only in a restricted part of England and in Ireland surveys of post-splenectomized patients have been performed. In Italy no common policy of patient care has yet been developed, and management of asplenia is mainly case or locally directed.

DETAILED DESCRIPTION:
People with asplenia have a high risk of serious infections, as the spleen is a reservoir of naive B and T cells and functions as a filter for antigens and capsulated bacteria in the blood. It also removes aged blood cells and Howell-Jolly's bodies from red blood cells.

The asplenia can be congenital, surgical and functional. Congenital asplenia is a condition associated with rare and poorly understood and studied syndromes. Surgical asplenia consists in the removal of the spleen for the management of some hematological or oncological diseases. Functional asplenia characterizes numerous hematological and non-hematological diseases; the most representative, among those hematological, is the sickle cell disease (SCD), among the non-hematological causes of functional asplenia, include several autoimmune diseases (e.g. Lupus, Sjogrens), inflammatory bowel disease (e.g. celiac disease, Crohn's disease, ulcerative rectocolitis ) and infiltrative diseases (e.g. amyloidosis, sarcoidosis).

Infections are the leading cause of death in individuals with asplenia, especially in children under the age of five . It has been shown that the integrity of the splenic function is necessary for the development and survival of IgM memory cells, a population of memory B cells of IgM isotype. These interesting data would explain the increased susceptibility to invasive infections sustained by capsulated bacteria in subjects with anatomical or functional asplenia, especially in the first years of life, in which there is a physiological and transient IgM memory deficit, supporting the common knowledge that the spleen represents a particular immunological environment that is fundamental for the removal of polysaccharide antigens and for the optimal antibody response.

In asplenic subjects, Streptococcus pneumoniae, Hemophilus influenzae and Neisseria meningitidis are the germs that most frequently cause invasive infections, such as bacteremia, sepsis and meningitis; therefore it is clear that prevention and immediate and aggressive treatment are the cornerstone of the correct management of this group of patients. Recently the new 13-valent conjugate vaccine against pneumococcus has been introduced and it is believed that this is a new and more effective strategy to reduce the infectious risk in these subjects; however, specific data on the population of asplenic subjects are lacking.

Recent studies and reports have shown a greater incidence of thrombotic complications in asplenic subjects, even if the rate of thrombotic events seems to be different between the different pathologies underlying the condition of asplenia. In fact, a large number of thrombotic events have been observed in splenectomized subjects for hereditary spherocytosis, for thalassemia, idiopathic thrombocytopenia purpura and other hematological diseases but the pathophysiological basis of these complications, the possible preventive treatments are not yet known. effective and optimal management of thrombotic events. Furthermore, preliminary data suggest a different susceptibility to infectious and thrombotic complications in the different forms of asplenia. If this is confirmed, the indications for antibiotic and antithrombotic prophylaxis, the timing of monitoring and the more or less aggressive management of complications, could vary in the different forms of asplenia.

Moreover, in Italy there are no shared and homogeneous indications on the prevention and treatment of short and long-term complications related to the condition of asplenia and their knowledge is still very limited among the medical staff. It has been shown that countries that have adopted shared measures for the management of these patients have achieved an improvement in the prevention of complications, through an increase vaccination coverage even among adults and the continuous information on possible risks related to the clinical condition. In fact, it often happens that patients do not respond to regular follow-up missing vaccination recalls and reducing over time all information about their health. This occurrence was considered one of the major risk factors for the development of serious complications in asplenic individuals .

The aim of the study is to retrospectively and prospectively assess a relatively large population of patients with asplenia in order to identify the rate of mortality and morbidity (infectious and thrombotic complications) developed by asplenic patients during the observation period.

ELIGIBILITY:
Inclusion Criteria:

* Adult and pediatric patients affected by asplenia

Exclusion Criteria:

* Medical history including all relevant clinical data required by the protocol not available

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients diagnosed with of any type of asplenia (congenital, surgical and functional) will be included in the study.
Sampling Method: Probability Sample
Enrollment: 1400 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2016-03-01 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
Identification of the causes of mortality and morbidity | 10 years
  The infectious and the thrombotic complication developed by asplenic patients during the observation period will be assessed

REFERENCES:
- [Background] Quinn CT, Rogers ZR, Buchanan GR. Survival of children with sickle cell disease. Blood. 2004 Jun 1;103(11):4023-7. doi: 10.1182/blood-2003-11-3758. Epub 2004 Feb 5. PMID 14764527
- [Background] Lee A, Thomas P, Cupidore L, Serjeant B, Serjeant G. Improved survival in homozygous sickle cell disease: lessons from a cohort study. BMJ. 1995 Dec 16;311(7020):1600-2. doi: 10.1136/bmj.311.7020.1600. PMID 8555802
- [Background] Gill FM, Sleeper LA, Weiner SJ, Brown AK, Bellevue R, Grover R, Pegelow CH, Vichinsky E. Clinical events in the first decade in a cohort of infants with sickle cell disease. Cooperative Study of Sickle Cell Disease. Blood. 1995 Jul 15;86(2):776-83. PMID 7606007
- [Background] Kruetzmann S, Rosado MM, Weber H, Germing U, Tournilhac O, Peter HH, Berner R, Peters A, Boehm T, Plebani A, Quinti I, Carsetti R. Human immunoglobulin M memory B cells controlling Streptococcus pneumoniae infections are generated in the spleen. J Exp Med. 2003 Apr 7;197(7):939-45. doi: 10.1084/jem.20022020. PMID 12682112
- [Background] Sullivan JL, Ochs HD, Schiffman G, Hammerschlag MR, Miser J, Vichinsky E, Wedgwood RJ. Immune response after splenectomy. Lancet. 1978 Jan 28;1(8057):178-81. doi: 10.1016/s0140-6736(78)90612-8. PMID 74605
- [Background] Pearson HA, Spencer RP, Cornelius EA. Functional asplenia in sickle-cell anemia. N Engl J Med. 1969 Oct 23;281(17):923-6. doi: 10.1056/NEJM196910232811703. No abstract available. PMID 5811425
- [Background] Hongeng S, Wilimas JA, Harris S, Day SW, Wang WC. Recurrent Streptococcus pneumoniae sepsis in children with sickle cell disease. J Pediatr. 1997 May;130(5):814-6. doi: 10.1016/s0022-3476(97)80026-1. PMID 9152293
- [Background] Casale M, Perrotta S. Splenectomy for hereditary spherocytosis: complete, partial or not at all? Expert Rev Hematol. 2011 Dec;4(6):627-35. doi: 10.1586/ehm.11.51. PMID 22077527
- [Background] Jais X, Ioos V, Jardim C, Sitbon O, Parent F, Hamid A, Fadel E, Dartevelle P, Simonneau G, Humbert M. Splenectomy and chronic thromboembolic pulmonary hypertension. Thorax. 2005 Dec;60(12):1031-4. doi: 10.1136/thx.2004.038083. Epub 2005 Aug 5. PMID 16085731
- [Background] Waghorn DJ. Overwhelming infection in asplenic patients: current best practice preventive measures are not being followed. J Clin Pathol. 2001 Mar;54(3):214-8. doi: 10.1136/jcp.54.3.214. PMID 11253134
- [Background] Hosea SW, Burch CG, Brown EJ, Berg RA, Frank MM. Impaired immune response of splenectomised patients to polyvalent pneumococcal vaccine. Lancet. 1981 Apr 11;1(8224):804-7. doi: 10.1016/s0140-6736(81)92681-7. PMID 6111673
- [Background] Wright J, Thomas P, Serjeant GR. Septicemia caused by Salmonella infection: an overlooked complication of sickle cell disease. J Pediatr. 1997 Mar;130(3):394-9. doi: 10.1016/s0022-3476(97)70201-4. PMID 9063414
- [Background] Taher AT, Musallam KM, Karimi M, El-Beshlawy A, Belhoul K, Daar S, Saned MS, El-Chafic AH, Fasulo MR, Cappellini MD. Overview on practices in thalassemia intermedia management aiming for lowering complication rates across a region of endemicity: the OPTIMAL CARE study. Blood. 2010 Mar 11;115(10):1886-92. doi: 10.1182/blood-2009-09-243154. Epub 2009 Dec 23. PMID 20032507